CLINICAL TRIAL: NCT05266989
Title: Effects of Transcranial Direct Current Stimulation on Brain Electrical Activity, Heart Rate Variability, and Dual-Task Performance in Healthy and Fibromyalgia Women
Brief Title: Effects of tDCS on People With Fibromyalgia
Status: Completed | Type: Observational
Sponsor: University of Extremadura (Other)
Collaborators: Ministerio de Asuntos Economicos y Transformación Digital, España (Unknown); Junta de Extremadura, España (Unknown)
Responsible Party: Principal Investigator, Narcis Gusi, Full Professor, University of Extremadura
Other Study IDs: 192/2021
Record Dates: First submitted 2022-02-01; First posted 2022-03-04 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Fibromyalgia
Keywords: Electroencephalography; EEG; Transcanial Stimulation; Strength
MeSH Terms: conditions — Fibromyalgia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fibromyalgia: All participants will randomly participate through three tDCS conditions (1mA, 2mA and sham)
  Interventions: Other: Transcranial Direct Current Stimulation
- Healthy Controls: All participants will randomly participate through three tDCS conditions (1mA, 2mA and sham)
  Interventions: Other: Transcranial Direct Current Stimulation

INTERVENTIONS:
Other: Transcranial Direct Current Stimulation — Non-invasive technique that modulates the excitability of the cortex by applying low-intensity current

SUMMARY:
People with fibromyalgia could experience physical and cognitive impairment as well as higher dual-task cost than healthy people when two tasks are performed simultaneously. Transcranial direct current stimulation is a promising non-pharmacological therapy. However, there is insufficient evidence about the intensities dose-response. Therefore, this protocol aims to 1) to compare the effectiveness and the impact of two tDCS intensities (1mA and 2mA) on cognitive, motor, brain functions, and cardiac autonomic modulation; 2) to study the impact of tDCS on the dual-task performance and creativity after applying tDCS in the dorsolateral prefrontal cortex. As hypotheses, a reduction of cognitive-motor interference in dual-task performance and also a modification in neurophysiological parameters, and an improvement in cardiac autonomic modulation are expected. Finally, no different effects are obtained depending on the intensity applied.

DETAILED DESCRIPTION:
Fibromyalgia is characterized by widespread pain and other associated symptoms, including stiffness, fatigue, non-recovery sleep, anxiety, or depression. On a physical level, people with FM frequently suffer from a sedentary state which reduces cardiovascular fitness and leads to mobility, strength and balance impairments. On a cognitive level, people with FM have often impaired cognitive functions such as memory, attention, processing speed, and executive functions. As a result of all of these symptoms, people with FM have a decreased performance in activities of daily living that are commonly presented as a simultaneous execution of two or more task at the same time (dual-task; DT).

To the knowledge of the investigators, no studies have focused on the application of transcranial direct current stimulation (tDCS) on the dorsolateral prefrontal cortex (DLPFC) to reduce the interference in DT performance. Furthermore, there are no studies that have studied the effects of different intensities of tDCS on DLPFC in people with FM in DT performance. Similarly, there are no studies that have focused on describing how neurophysiological variables may be modified in people with FM during DT performance. Therefore, it seems interesting to know how tDCS can influence these types of variables in order to improve the quality of life of this population and to open new frontiers for research.

The hypotheses that are proposed for this study are as follows: a) the application of tDCS will improve physical performance in physical variables that will be measured through balance and strength tasks; b) the application of tDCS will improve performance on neurophysiological variables that will be measured through brain electrical activity and HRV; c) the application of tDCS will improve performance in DT conditions as well as in creativity tasks; d) tDCS will have different effects depending on the variability of fibromyalgia symptoms presented (pain, sleep problems and depression); e) no significant effects on the variables would be expected depending on the type of tDCS intensity applied.

At this point, the main objectives of this protocol are: 1) to compare the effectiveness and the impact of two tDCS intensities (1mA and 2mA) on neurophysiological variables, cognitive, and motor functions; 2) to study the impact of tDCS on the dual-task performance and creativity after applying tDCS in dorsolateral prefrontal cortex.

ELIGIBILITY:
Inclusion Criteria:

* Be able to communicate with the research staff
* Have read, understood, and signed the informed consent form

Exclusion Criteria:

* Physiatric or neurological disorders
* Pharmacological treatment for anxiety or depression
* Substance abuse or dependence
* Contraindication for physical effort
* Difficulty in maintaining balance
* Leg injury that interferes with flexion and extension of the knee
* Being pregnant

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy and fibromyalgia women living in Caceres (Spain) and the surrounding area
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
Degree of change in electroencephalography (EEG) between pre and post tDCS session | Once before and after each tDCS session
  The Enobio instrument (Neuroelectrics) and Neuroelectrics instrument driver software (NIC1) will be used to record EEG. Theta, alpha and beta power spectrums will be extracted from a 5 minute recording.
Degree of change in heart rate variability (HRV) between pre and post tDCS session | Once before and after each tDCS session
  The Enobio instrument (Neuroelectrics) and Neuroelectrics instrument driver software (NIC1) will be used to record HRV. Time domain (SDNN, RMSSD, RR-interval and pNN50), frequency domain (LFnu, HFnu, LF/HF and total power) and non-linear measures (SampEn, SD1 and SD2) will be extracted from a 5 minute recording.
Degree of change in balance between pre and post tDCS session | Once before and after each tDCS session
  The tests will be static position with eyes open and static position with eyes closed. The test will be performed on a Kistler force platform.
Degree of change in strength between pre and post tDCS session | Once before and after each tDCS session
  The execution of the test consists of performing a concentric contraction of knee flexion and extension six times consecutively and without pause between repetitions at a speed of 60 /s and in a range of movement from 0 to 90 degrees, being 0 full extension and 90 flexion. The test will be performed on the isokinetic dynamometer Multi-Joint 3, Biodex Medical Sistems.
Degree of change in balance, under dual-task condition, between pre and post tDCS session | Once before and after each tDCS session
  Participants will simultaneously perform the balance test (static position with eyes open and static position with eyes closed) and a cognitive task. The cognitive task will consist of two-by-two substractions from a number greater than 100.
Degree of change in strenght, under dual-task condition, between pre and post tDCS session | Once before and after each tDCS session
  Participants will simultaneously perform the strenght test (conducting a concentric contraction of knee flexion and extension six times consecutively and without pause between repetitions at a speed of 60 /s and in a range of movement from 0 to 90 degrees, being 0 full extension and 90 flexion) and a cognitive task. The cognitive task will consist of two-by-two substractions from a number greater than 100.

SECONDARY OUTCOMES:
Socio-demographic information | At week 1
  Age, level of education, injuries, or falls in the last few months, as well as other health related information, will be asked.
Physical activity level | At week 1
  International Physical activity Questionnaire (IPAQ): results can be reported in categories (low activity levels, moderate activity levels or high activity levels) or as a continuous variable (MET minutes a week). MET minutes represent the amount of energy expended carrying out physical activity. Scoring a low level of physical activity on the IPAQ means that you are not meeting any of the criteria for either moderate or high levels of physical activity.
Impact of the disease | At week 1
  Fibromialgia Impact Questionnaire Revised (FIQ-R): the minimum score is 0 and the maximum is 100, corresponding to the worst overall symptom impact.
Fear of falling | At week 1
  Falls Efficacy Scale International (FES-I): the minimum score is 16 and the maximum is 64. The higher the score, the greater the fear of falling.
Health-related quality of life | At week 1
  EuroQol- 5 dimensions- 5 levels (EQ-5D-5L) (range 0 to 100 with higher values corresponding to better health status).
Sleep Quality | At week 1
  Pittsburg Sleep Quality Index (PSQI) (range 0 to 21, with higher score referring to worse sleep quality).
Cognitive Impairment | At week 1
  Montreal Cognitive Assessment (MoCA) (range 0 to 35 with higher values corresponding to better cognitive function).
Degree of change in sensations related to tDCS | Once after the tDCS sessions
  Survey of sensations related to tDCS
Bioelectrical impedance analysis | At week 1
  Body composition will be measured with the Tanita BC-418 Body Composition Analyzer
Height (meters) | At week 1
  Using a SECA 285 model.

CONTACTS AND LOCATIONS:
Overall Officials: Narcis Gusi, Study Director — Universidad de Extremadura
Locations (1):
- Facultad de Ciencias del Deporte, Cáceres, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing will be evaluated upon reasonable request by the research group.